CLINICAL TRIAL: NCT00097916
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Memantine in Non-Institutionalized Agitated Patients With Moderate to Severe Alzheimer's Disease
Brief Title: An Evaluation of the Safety and Efficacy of Memantine in Agitated Patients With Moderate to Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEM-MD-23
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Alzheimer's Disease
Keywords: memantine HCl; Dementia; Agitation; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychomotor Agitation | interventions — Memantine

INTERVENTIONS:
Drug: memantine HCl

SUMMARY:
About 65% of patients with severe Alzheimer's Disease (AD) will have symptoms of agitation. There are drawbacks associated with the currently available therapeutic interventions for agitation associated with Alzheimer's Disease. In a recent trial, in the group of patients with moderate to severe AD treated with memantine, there were fewer incidences of agitation. It is hypothesized that memantine will be effective in reducing the symptoms of agitation associated with moderate to severe Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to Severe Alzheimer's Disease with a score greater than or equal to 4 on agitation/aggression domain of NPI
* Stable dose of donepezil for 3 months

Exclusion Criteria:

* Other evidence of psychiatric disorders
* Oncologic diagnosis
* Clinically significant gastrointestinal, renal, hepatic, endocrine or cardiovascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory

SECONDARY OUTCOMES:
Cohen Mansfield Agitation Inventory
Clinical Global Impression Scale
ADCS-ADL
Agitation/aggression domain of Neuropsychiatric Inventory (NPI)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - The Forves Norris MDA/ALS Research Center, San Francisco, California
  - Coastal Communities Hospital, Westminster, California
  - Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Berma Research Group, Hialeah, Florida
  - Baumel-Eisner Neuromedical Institute, Miami, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Geriatric Medicine, Honolulu, Hawaii
  - The Memory Clinic, Bennington, Vermont
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia